CLINICAL TRIAL: NCT01414023
Title: Assessing the Effects of a Neurobehavioral Intervention on Symptoms of Obsessive Compulsive Disorder
Acronym: CCT-OC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BU-2487; NCT01414023 (Registry Identifier: Clinical Trials)
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Obsessive Compulsive Disorder
Keywords: High OCI-R scores
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CCT (Experimental): Cognitive Control Training - Pace Auditory Serial Addition Task (PASAT;(Gronwall, 1977): A computer version of the PASAT will be used to measure sustained attention and working memory. Participants are asked to add serially presented numbers. Attention Control Intervention (Wells, 2000): This task involves training individuals to attend differentially to multiple auditory sources (e.g., by counting tones, discriminating the location of tones, and moving their attention between auditory sources for a prolonged period).
  Interventions: Behavioral: Cognitive Control Training
- PVT (Placebo Comparator): Peripheral Vision Task (PVT; C. Moore, personal communication): This task serves as a non-active control condition which does not target the brain regions influenced by the Wells and PASAT tasks. Participants focus on the placement of dots on a computer screen in this task while listening to a tone.
  Interventions: Behavioral: Peripheral Vision Task

INTERVENTIONS:
Behavioral: Cognitive Control Training — Pace Auditory Serial Addition Task (PASAT;(Gronwall, 1977): A computer version of the PASAT will be used to measure sustained attention and working memory. Participants are asked to add serially presented numbers. Attention Control Intervention (Wells, 2000): This task involves training individuals to attend differentially to multiple auditory sources (e.g., by counting tones, discriminating the location of tones, and moving their attention between auditory sources for a prolonged period).
  Arms: CCT
Behavioral: Peripheral Vision Task — Peripheral Vision Task (PVT; C. Moore, personal communication): This task serves as a non-active control condition which does not target the brain regions influenced by the Wells and PASAT tasks. Participants focus on the placement of dots on a computer screen in this task while listening to a tone.
  Arms: PVT

SUMMARY:
This experiment will examine if the use of computerized tasks that train individuals to control their attention more effectively will predict individual differences in obsessive-compulsive symptoms, rumination and BDNF change. After giving consent, filling out self-report forms, and giving blood for the BDNF test, 80 participants will be randomized to Cognitive Control Training (CCT) or Peripheral Vision Task (PVT) (described below) which will be administered three times over a two week period. At the third visit, participants will also complete an anagram task and repeat the blood draw for BDNF testing. The investigators hypothesize that computerized tasks that train individuals to control their attention more effectively will reduce Obsessive Compulsive (OC) symptoms. Additionally, individuals training in CCT will show increased ability to disengage from unattainable goals as assessed by responses to an unsolvable anagram task. Finally, individuals training in CCT will show a greater increase in BDNF levels as compared to individuals training in PVT.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-65 years
* OCI-R total score ≥ 16
* Ability to read and provide informed consent.
* Familiarity with a computer keyboard and mouse.

Exclusion Criteria:

* BDI-II suicidality score of > 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
OCI-R scores | up to two weeks
  3 times over a two week period

SECONDARY OUTCOMES:
BDNF serum levels | up to two weeks
  Two times over a two week period

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States